CLINICAL TRIAL: NCT03000751
Title: CT Dose Optimization and Standardization Endeavor (DOSE) Collaboratory
Brief Title: CT DOSE Collaboratory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Davis (Other); University Hospital, Basel, Switzerland (Other); Center for Diagnostic Imaging (Other); Community Health Network (Other); Children's Mercy Hospital Kansas City (Other); City of Hope Medical Center (Other); Albert Einstein Healthcare Network (Other); Universität Duisburg-Essen (Other); East Texas Medical Center Regional Healthcare System (Other); Emory University (Other); Henry Ford Health System (Other); Huntsville Hospital Health System (Other); Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other); Mount Sinai Hospital, New York (Other); Maastricht University Medical Center (Other); Olive View-UCLA Education & Research Institute (Other); Oxford University Hospitals NHS Trust (Other); San Francisco VA Health Care System (U.S. Federal Agency); St. Joseph Hospital of Orange (Other); St. Luke's International Hospital, Japan (Other); University of Virginia (Other); University of California, Irvine (Other); University of California, San Diego (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: RSB-181191; R01CA181191 (NIH)
Record Dates: First submitted 2016-12-12; First posted 2016-12-22 (Estimated); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Ionizing Radiation Exposure; Quality Improvement
Keywords: CT scan; CT exam; ionizing radiation; medical imaging; cat scan; radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Track A (Active Comparator): Simple Audit Report; In-Person Meeting (timed to coincide with the multi-component intervention); Multi-Component Intervention
  Interventions: Other: Simple Audit Report; Other: Multi-Component Intervention; Other: In-Person Meeting
- Track B (Active Comparator): In-Person Meeting (timed to coincide with the simple audit report); Simple Audit Report; Multi-Component Intervention
  Interventions: Other: Simple Audit Report; Other: Multi-Component Intervention; Other: In-Person Meeting
- Track C (Other): Simple Audit Report; Multi-Component Intervention
  Interventions: Other: Simple Audit Report; Other: Multi-Component Intervention

INTERVENTIONS:
Other: Simple Audit Report — The simple audit provides comparison and feedback on radiation doses.
Other: Multi-Component Intervention — The multi-component intervention gives tailored feedback on needed changes plus guidance using quality improvement methods that facilitate organizational change. Provides access to experts, detailed audit, collaborative calls, and site visits (as needed).
Other: In-Person Meeting — Collaborator meeting with an emphasis on quality improvement.
  Arms: Track A; Track B

SUMMARY:
This is a pragmatic stepped-wedge cluster randomized controlled trial to explore variation in doses used for diagnostic CT by pooling radiation dose data across diverse healthcare delivery systems.

To compare different strategies for lowering and optimizing dose and identify the barriers and facilitators to implementing successful dose optimization strategies and standardizing practice.

DETAILED DESCRIPTION:
The investigators are using a stepped-wedge cluster randomized controlled trial, collecting radiation dose information on CT from across all collaborating health care facilities, and leading several different interventions to optimize dose across facilities. In addition to collecting the CT radiation dose data, and using these results to provide feedback to the collaborating health care facilities, they will be conducting surveys of several individuals at each site, including key informants, such as lead radiologists, technologists, and medical physicist, and radiology administrators.

They will compare and identify facilitators and barriers (assessed through surveys of participating facilities) associated with successful and failed implementation of dose optimization.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic CT scans of the head, chest, and/or abdomen/pelvis performed within the study period

Exclusion Criteria:

* non-diagnostic scans that are not of the head, chest, and/or abdomen/pelvis

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 864080 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Smith-Bindman, MD, Principal Investigator — University of California, San Francisco; Judy Yee, MD, Principal Investigator — San Francisco Veterans Administration; Tom Nelson, PhD, Principal Investigator — University of California, San Diego; Tony Seibert, PhD, Principal Investigator — University of California, Davis; Mayil Krishnam, MD, Principal Investigator — University of California, Irvine; Michael Flynn, PhD, Principal Investigator — Henry Ford Health System; Mary Cocker, MSc, Csci, Principal Investigator — Oxford University Hospitals NHS Trust; William Boswell, MD, Principal Investigator — City of Hope Medical Center; Sebastian Schindera, MD, Principal Investigator — University Hospital of Basel; Erin Bell, MHP, Principal Investigator — Community Health Network; Phuong-Anh Duong, MD, Principal Investigator — Emory University; Nima Kasraie, PhD, MSc, Principal Investigator — Children's Mercy Hospital Kansas City; Pavlina Pike, PhD, Principal Investigator — Huntsville Hospital; Luisa Cervantes, MD, Principal Investigator — Nicklaus Children's Hospital f/k/a Miami Children's Hospital; Joachim Wildberger, PhD, Principal Investigator — Maastricht University Medical Center; Michael Forsting, MD, Principal Investigator — University of Duisburg-Essen; Fady Kassem, PhD, Principal Investigator — St. Joseph Hospital of Orange; Darrell Fendrick, CT, Principal Investigator — East Texas Medical Center; Sugoto Mukherjee, MD, Principal Investigator — University of Virginia Health System; Brad Delman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Jodi Roehm, Principal Investigator — Center for Diagnostic Imaging; Anokh Pahwa, MD, Principal Investigator — Olive View - UCLA; Ryan Lee, MD, MBA, Principal Investigator — Einstein Medical Center; Jay Starkey, MD, Principal Investigator — St. Luke's International Hospital, Tokyo; Diana Miglioretti, PhD, Principal Investigator — University of California, Davis; Saravanabavaan Suntharalingam, MD, Principal Investigator — University of Duisburg-Essen; Sara Lewis, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Solberg LI. Improving medical practice: a conceptual framework. Ann Fam Med. 2007 May-Jun;5(3):251-6. doi: 10.1370/afm.666. PMID 17548853
- [Background] Solberg LI, Asche SE, Margolis KL, Whitebird RR. Measuring an organization's ability to manage change: the change process capability questionnaire and its use for improving depression care. Am J Med Qual. 2008 May-Jun;23(3):193-200. doi: 10.1177/1062860608314942. PMID 18539980
- [Background] Schindera ST, Treier R, von Allmen G, Nauer C, Trueb PR, Vock P, Szucs-Farkas Z. An education and training programme for radiological institutes: impact on the reduction of the CT radiation dose. Eur Radiol. 2011 Oct;21(10):2039-45. doi: 10.1007/s00330-011-2168-5. Epub 2011 May 31. PMID 21626359
- [Background] Keegan J, Miglioretti DL, Gould R, Donnelly LF, Wilson ND, Smith-Bindman R. Radiation dose metrics in CT: assessing dose using the National Quality Forum CT patient safety measure. J Am Coll Radiol. 2014 Mar;11(3):309-15. doi: 10.1016/j.jacr.2013.10.009. PMID 24589407
- [Background] Miglioretti DL, Zhang Y, Johnson E, Lee C, Morin RL, Vanneman N, Smith-Bindman R. Personalized technologist dose audit feedback for reducing patient radiation exposure from CT. J Am Coll Radiol. 2014 Mar;11(3):300-8. doi: 10.1016/j.jacr.2013.10.017. PMID 24589406
- [Background] Pearce MS, Salotti JA, Little MP, McHugh K, Lee C, Kim KP, Howe NL, Ronckers CM, Rajaraman P, Sir Craft AW, Parker L, Berrington de Gonzalez A. Radiation exposure from CT scans in childhood and subsequent risk of leukaemia and brain tumours: a retrospective cohort study. Lancet. 2012 Aug 4;380(9840):499-505. doi: 10.1016/S0140-6736(12)60815-0. Epub 2012 Jun 7. PMID 22681860
- [Background] Mathews JD, Forsythe AV, Brady Z, Butler MW, Goergen SK, Byrnes GB, Giles GG, Wallace AB, Anderson PR, Guiver TA, McGale P, Cain TM, Dowty JG, Bickerstaffe AC, Darby SC. Cancer risk in 680,000 people exposed to computed tomography scans in childhood or adolescence: data linkage study of 11 million Australians. BMJ. 2013 May 21;346:f2360. doi: 10.1136/bmj.f2360. PMID 23694687
- [Background] Conference of Radiation Control Program Directors. Nationwide evaluation of x-ray trends (NEXT): Tabulation and graphical summary of 2000 survey of computed tomography . Frankfort, KY2007.
- [Background] Bhargavan M, Sunshine JH. Utilization of radiology services in the United States: levels and trends in modalities, regions, and populations. Radiology. 2005 Mar;234(3):824-32. doi: 10.1148/radiol.2343031536. Epub 2005 Jan 28. PMID 15681686
- [Background] Smith-Bindman R, Miglioretti DL, Larson EB. Rising use of diagnostic medical imaging in a large integrated health system. Health Aff (Millwood). 2008 Nov-Dec;27(6):1491-502. doi: 10.1377/hlthaff.27.6.1491. PMID 18997204
- [Background] Baker LC, Atlas SW, Afendulis CC. Expanded use of imaging technology and the challenge of measuring value. Health Aff (Millwood). 2008 Nov-Dec;27(6):1467-78. doi: 10.1377/hlthaff.27.6.1467. PMID 18997202
- [Background] Medicare Payment Advisory Commission. A Data Book: Healthcare Spending and the Medicare Program, June 2010.
- [Background] Levin DC, Rao VM, Parker L, Frangos AJ, Sunshine JH. Bending the curve: the recent marked slowdown in growth of noninvasive diagnostic imaging. AJR Am J Roentgenol. 2011 Jan;196(1):W25-9. doi: 10.2214/AJR.10.4835. PMID 21178027
- [Background] Smith-Bindman R, Miglioretti DL, Johnson E, Lee C, Feigelson HS, Flynn M, Greenlee RT, Kruger RL, Hornbrook MC, Roblin D, Solberg LI, Vanneman N, Weinmann S, Williams AE. Use of diagnostic imaging studies and associated radiation exposure for patients enrolled in large integrated health care systems, 1996-2010. JAMA. 2012 Jun 13;307(22):2400-9. doi: 10.1001/jama.2012.5960. PMID 22692172
- [Background] Mettler FA Jr, Huda W, Yoshizumi TT, Mahesh M. Effective doses in radiology and diagnostic nuclear medicine: a catalog. Radiology. 2008 Jul;248(1):254-63. doi: 10.1148/radiol.2481071451. PMID 18566177
- [Background] National Council on Radiation Protection and Measurements. NCRP Report No. 93, Ionizing Radiation Exposure of the Population of the United States. 1987
- [Background] National Council on Radiation Protection and Measurements. NCRP Report No 160, Ionizing Radiation Exposure of the Population of the United States, press release available , full report soon to be released; 2009
- [Background] Pierce DA, Preston DL. Radiation-related cancer risks at low doses among atomic bomb survivors. Radiat Res. 2000 Aug;154(2):178-86. doi: 10.1667/0033-7587(2000)154[0178:rrcral]2.0.co;2. PMID 10931690
- [Background] Preston DL, Ron E, Tokuoka S, Funamoto S, Nishi N, Soda M, Mabuchi K, Kodama K. Solid cancer incidence in atomic bomb survivors: 1958-1998. Radiat Res. 2007 Jul;168(1):1-64. doi: 10.1667/RR0763.1. PMID 17722996
- [Background] Brenner DJ, Doll R, Goodhead DT, Hall EJ, Land CE, Little JB, Lubin JH, Preston DL, Preston RJ, Puskin JS, Ron E, Sachs RK, Samet JM, Setlow RB, Zaider M. Cancer risks attributable to low doses of ionizing radiation: assessing what we really know. Proc Natl Acad Sci U S A. 2003 Nov 25;100(24):13761-6. doi: 10.1073/pnas.2235592100. Epub 2003 Nov 10. PMID 14610281
- [Background] Board of Radiation Effects Research Division on Earth and Life Sciences National Research Council of the National Academies. Health Risks from Exposure to Low Levels of Ionizing Radiation: BEIR VII Phase 2 Washington, D.C.: The National Academies Press; 2006.
- [Background] Boutis K, Cogollo W, Fischer J, Freedman SB, Ben David G, Thomas KE. Parental knowledge of potential cancer risks from exposure to computed tomography. Pediatrics. 2013 Aug;132(2):305-11. doi: 10.1542/peds.2013-0378. Epub 2013 Jul 8. PMID 23837174
- [Background] Hertz-Picciotto I. Breast Cancer and the Environment: A Life Course Approach. Dec 2011 2011.
- [Background] Berrington de Gonzalez A, Mahesh M, Kim KP, Bhargavan M, Lewis R, Mettler F, Land C. Projected cancer risks from computed tomographic scans performed in the United States in 2007. Arch Intern Med. 2009 Dec 14;169(22):2071-7. doi: 10.1001/archinternmed.2009.440. PMID 20008689
- [Background] Berrington de Gonzalez A, Darby S. Risk of cancer from diagnostic X-rays: estimates for the UK and 14 other countries. Lancet. 2004 Jan 31;363(9406):345-51. doi: 10.1016/S0140-6736(04)15433-0. PMID 15070562
- [Background] Smith-Bindman R, Lipson J, Marcus R, Kim KP, Mahesh M, Gould R, Berrington de Gonzalez A, Miglioretti DL. Radiation dose associated with common computed tomography examinations and the associated lifetime attributable risk of cancer. Arch Intern Med. 2009 Dec 14;169(22):2078-86. doi: 10.1001/archinternmed.2009.427. PMID 20008690
- [Background] Rydberg J, Buckwalter KA, Caldemeyer KS, Phillips MD, Conces DJ Jr, Aisen AM, Persohn SA, Kopecky KK. Multisection CT: scanning techniques and clinical applications. Radiographics. 2000 Nov-Dec;20(6):1787-806. doi: 10.1148/radiographics.20.6.g00nv071787. PMID 11112829
- [Background] Halpern EJ. Triple-rule-out CT angiography for evaluation of acute chest pain and possible acute coronary syndrome. Radiology. 2009 Aug;252(2):332-45. doi: 10.1148/radiol.2522082335. PMID 19703877
- [Background] Sommer WH, Schenzle JC, Becker CR, Nikolaou K, Graser A, Michalski G, Neumaier K, Reiser MF, Johnson TR. Saving dose in triple-rule-out computed tomography examination using a high-pitch dual spiral technique. Invest Radiol. 2010 Feb;45(2):64-71. doi: 10.1097/RLI.0b013e3181c15842. PMID 20027121
- [Background] Foley WD, Mallisee TA, Hohenwalter MD, Wilson CR, Quiroz FA, Taylor AJ. Multiphase hepatic CT with a multirow detector CT scanner. AJR Am J Roentgenol. 2000 Sep;175(3):679-85. doi: 10.2214/ajr.175.3.1750679. PMID 10954450
- [Background] Roberts HC, Roberts TP, Smith WS, Lee TJ, Fischbein NJ, Dillon WP. Multisection dynamic CT perfusion for acute cerebral ischemia: the "toggling-table" technique. AJNR Am J Neuroradiol. 2001 Jun-Jul;22(6):1077-80. PMID 11415901
- [Background] Hoeffner EG, Case I, Jain R, Gujar SK, Shah GV, Deveikis JP, Carlos RC, Thompson BG, Harrigan MR, Mukherji SK. Cerebral perfusion CT: technique and clinical applications. Radiology. 2004 Jun;231(3):632-44. doi: 10.1148/radiol.2313021488. Epub 2004 Apr 29. PMID 15118110
- [Background] Smith AB, Dillon WP, Lau BC, Gould R, Verdun FR, Lopez EB, Wintermark M. Radiation dose reduction strategy for CT protocols: successful implementation in neuroradiology section. Radiology. 2008 May;247(2):499-506. doi: 10.1148/radiol.2472071054. Epub 2008 Mar 27. PMID 18372456
- [Background] Caoili EM, Cohan RH, Ellis JH, Dillman J, Schipper MJ, Francis IR. Medical decision making regarding computed tomographic radiation dose and associated risk: the patient's perspective. Arch Intern Med. 2009 Jun 8;169(11):1069-71. doi: 10.1001/archinternmed.2009.139. No abstract available. PMID 19506177
- [Background] Smith-Bindman R. Is computed tomography safe? N Engl J Med. 2010 Jul 1;363(1):1-4. doi: 10.1056/NEJMp1002530. Epub 2010 Jun 23. No abstract available. PMID 20573919
- [Background] Duncan JR, Evens RG. Using information to optimize medical outcomes. JAMA. 2009 Jun 10;301(22):2383-5. doi: 10.1001/jama.2009.827. No abstract available. PMID 19509387
- [Background] Poletti PA, Platon A, Rutschmann OT, Schmidlin FR, Iselin CE, Becker CD. Low-dose versus standard-dose CT protocol in patients with clinically suspected renal colic. AJR Am J Roentgenol. 2007 Apr;188(4):927-33. doi: 10.2214/AJR.06.0793. PMID 17377025
- [Background] Radiation protection 118 : referral guidelines for imaging. Luxembourg European Commission, Directorate- General for the Environment; 2001
- [Background] U.S. Food and Drug Administration. FDA White Paper: Initiative to Reduce Unnecessary Radiation Exposure from Medical Imaging. 2010; http://www.fda.gov/Radiation- EmittingProducts/RadiationSafety/RadiationDoseReduction/ucm199994.htm.
- [Background] US Food and Drug Administration. Safety Investigation of CT Brain Perfusion Scans: Update 11/9/2010. 2009
- [Background] Bogdanich W. After stroke scans, patients face serious risk. New York TImes. July 31, 2010, 2010.
- [Background] Bogdanich W. Listing of articles published in the NY TImes over the last year in the 'Radiation Boom' series by Walt Bogdanich examine issues arising from the increasing use of medical radiation and the new technologies that deliver it. . http://topics.nytimes.com/top/news/us/series/radiation_boom/index.html?ref=health.
- [Background] The US House of Representatives, Energy and Commerce Committee, Subcommittee on Health held a hearing entitled
- [Background] Brody AS, Frush DP, Huda W, Brent RL; American Academy of Pediatrics Section on Radiology. Radiation risk to children from computed tomography. Pediatrics. 2007 Sep;120(3):677-82. doi: 10.1542/peds.2007-1910. PMID 17766543
- [Background] UK National Health Program Department of Health. The Ionising Radiation (Medical Exposure) Regulations 2000 (together with notes on good practice). 2007, http://www.dh.gov.uk/en/Publicationsandstatistics/Publications/PublicationsPolicyAndGuidance/DH_4007957, accessed January 15, 2011
- [Background] Wall BF. Diagnostic reference levels--the way forward. Br J Radiol. 2001 Sep;74(885):785-8. doi: 10.1259/bjr.74.885.740785. No abstract available. PMID 11560825
- [Background] 1990 Recommendations of the International Commission on Radiological Protection. Ann ICRP. 1991;21(1-3):1-201. No abstract available. PMID 2053748
- [Background] Radiological protection and safety in medicine. A report of the International Commission on Radiological Protection. Ann ICRP. 1996;26(2):1-47. No abstract available. PMID 8911634
- [Background] Seeram E, Brennan PC. Diagnostic reference levels in radiology. Radiol Technol. 2006 May-Jun;77(5):373-84; quiz 385-7. No abstract available. PMID 16709686
- [Background] Amis ES Jr, Butler PF, Applegate KE, Birnbaum SB, Brateman LF, Hevezi JM, Mettler FA, Morin RL, Pentecost MJ, Smith GG, Strauss KJ, Zeman RK; American College of Radiology. American College of Radiology white paper on radiation dose in medicine. J Am Coll Radiol. 2007 May;4(5):272-84. doi: 10.1016/j.jacr.2007.03.002. PMID 17467608
- [Background] Smith-Bindman R. Environmental causes of breast cancer and radiation from medical imaging: findings from the Institute of Medicine report. Arch Intern Med. 2012 Jul 9;172(13):1023-7. doi: 10.1001/archinternmed.2012.2329. PMID 22688684
- [Background] Center for Medicare and Medicaid Services. Section 135(b)of the Medicare Improvements for Patients and Providers Act of 2008 (MIPPA) mandates an Appropriate Use of Imaging Services demonstration project. The goal of the demonstration is to collect data regarding physician use of advanced diagnostic imaging services to determine the appropriateness of services in relation to established criteria and physician peers. 2010; http://www.cms.gov/demoprojectsevalrpts/md/itemdetail.asp?itemid=CMS1222075.
- [Background] The Joint Commission Sentinel Event Alert System. 2011; http://www.jointcommission.org/assets/1/18/SEA_471.PDF.
- [Background] Image Gently. 2009. http://www.pedrad.org/associations/5364/ig/index.cfm?page=369. Accessed Feb 13, 2009.
- [Background] Catalano C, Francone M, Ascarelli A, Mangia M, Iacucci I, Passariello R. Optimizing radiation dose and image quality. Eur Radiol. 2007 Dec;17 Suppl 6:F26-32. doi: 10.1007/s10406-007-0225-6. PMID 18376454
- [Background] Lee CI, Haims AH, Monico EP, Brink JA, Forman HP. Diagnostic CT scans: assessment of patient, physician, and radiologist awareness of radiation dose and possible risks. Radiology. 2004 May;231(2):393-8. doi: 10.1148/radiol.2312030767. Epub 2004 Mar 18. PMID 15031431
- [Background] Damschroder LJ, Banaszak-Holl J, Kowalski CP, Forman J, Saint S, Krein SL. The role of the champion in infection prevention: results from a multisite qualitative study. Qual Saf Health Care. 2009 Dec;18(6):434-40. doi: 10.1136/qshc.2009.034199. PMID 19955453
- [Background] Aarons G, Horowitz J, Dlugosz L, Ehrhart M. The role of organizational processes in dissemination and implementation researach. In: Brownson RC, Colditz GA, Proctor EK, eds. Dissemination and Implementation Research in Health: Translating Science to Practice. New York: Oxford University Press, Inc.; 2012:
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Solberg LI, Asche SE, Margolis KL, Whitebird RR, Trangle MA, Wineman AP. Relationship between the presence of practice systems and the quality of care for depression. Am J Med Qual. 2008 Nov-Dec;23(6):420-6. doi: 10.1177/1062860608324547. PMID 19001099
- [Background] Glasgow RE, Klesges LM, Dzewaltowski DA, Estabrooks PA, Vogt TM. Evaluating the impact of health promotion programs: using the RE-AIM framework to form summary measures for decision making involving complex issues. Health Educ Res. 2006 Oct;21(5):688-94. doi: 10.1093/her/cyl081. Epub 2006 Aug 31. PMID 16945984
- [Background] Fortney J, Enderle M, McDougall S, Clothier J, Otero J, Altman L, Curran G. Implementation outcomes of evidence-based quality improvement for depression in VA community based outpatient clinics. Implement Sci. 2012 Apr 11;7:30. doi: 10.1186/1748-5908-7-30. PMID 22494428
- [Background] Glasgow RE. RE-AIMing research for application: ways to improve evidence for family medicine. J Am Board Fam Med. 2006 Jan-Feb;19(1):11-9. doi: 10.3122/jabfm.19.1.11. PMID 16492000
- [Background] Cho RC, Chu P, Smith-Bindman R. Second trimester prenatal ultrasound for the detection of pregnancies at increased risk of Trisomy 18 based on serum screening. Prenat Diagn. 2009 Feb;29(2):129-39. doi: 10.1002/pd.2166. PMID 19142904
- [Background] Haggstrom DA, Quale C, Smith-Bindman R. Differences in the quality of breast cancer care among vulnerable populations. Cancer. 2005 Dec 1;104(11):2347-58. doi: 10.1002/cncr.21443. PMID 16211547
- [Background] Kagay CR, Quale C, Smith-Bindman R. Screening mammography in the American elderly. Am J Prev Med. 2006 Aug;31(2):142-9. doi: 10.1016/j.amepre.2006.03.029. PMID 16829331
- [Background] Kerlikowske K, Smith-Bindman R, Abraham LA, Lehman CD, Yankaskas BC, Ballard-Barbash R, Barlow WE, Voeks JH, Geller BM, Carney PA, Sickles EA. Breast cancer yield for screening mammographic examinations with recommendation for short-interval follow-up. Radiology. 2005 Mar;234(3):684-92. doi: 10.1148/radiol.2343031976. PMID 15734926
- [Background] Levine D, Brown DL, Andreotti RF, Benacerraf B, Benson CB, Brewster WR, Coleman B, DePriest P, Doubilet PM, Goldstein SR, Hamper UM, Hecht JL, Horrow M, Hur HC, Marnach M, Patel MD, Platt LD, Puscheck E, Smith-Bindman R; Society of Radiologists in Ultrasound. Management of asymptomatic ovarian and other adnexal cysts imaged at US Society of Radiologists in Ultrasound consensus conference statement. Ultrasound Q. 2010 Sep;26(3):121-31. doi: 10.1097/RUQ.0b013e3181f09099. PMID 20823748
- [Background] Miglioretti DL, Smith-Bindman R, Abraham L, Brenner RJ, Carney PA, Bowles EJ, Buist DS, Elmore JG. Radiologist characteristics associated with interpretive performance of diagnostic mammography. J Natl Cancer Inst. 2007 Dec 19;99(24):1854-63. doi: 10.1093/jnci/djm238. Epub 2007 Dec 11. PMID 18073379
- [Background] Schueler K, Chu P, Smith-Bindman R. "Racial Differences in the Use of Mammography:" A Meta-analytical Review of Literature Describing Economic, Social, and Cultural Reasons for Variation in Use of Mammography". Submitted. 2005
- [Background] Sickles EA, Miglioretti DL, Ballard-Barbash R, Geller BM, Leung JW, Rosenberg RD, Smith-Bindman R, Yankaskas BC. Performance benchmarks for diagnostic mammography. Radiology. 2005 Jun;235(3):775-90. doi: 10.1148/radiol.2353040738. PMID 15914475
- [Background] Smith-Bindman R, Ballard-Barbash R, Miglioretti DL, Patnick J, Kerlikowske K. Comparing the performance of mammography screening in the USA and the UK. J Med Screen. 2005;12(1):50-4. doi: 10.1258/0969141053279130. PMID 15814020
- [Background] Smith-Bindman R, Chu P, Bacchetti P, Waters JJ, Mutton D, Alberman E. Prenatal screening for Down syndrome in England and Wales and population-based birth outcomes. Am J Obstet Gynecol. 2003 Oct;189(4):980-5. doi: 10.1067/s0002-9378(03)00721-x. PMID 14586339
- [Background] Smith-Bindman R, Chu P, Goldberg JD. Second trimester prenatal ultrasound for the detection of pregnancies at increased risk of Down syndrome. Prenat Diagn. 2007 Jun;27(6):535-44. doi: 10.1002/pd.1725. PMID 17367102
- [Background] Smith-Bindman R, Chu P, Miglioretti DL, Quale C, Rosenberg RD, Cutter G, Geller B, Bacchetti P, Sickles EA, Kerlikowske K. Physician predictors of mammographic accuracy. J Natl Cancer Inst. 2005 Mar 2;97(5):358-67. doi: 10.1093/jnci/dji060. PMID 15741572
- [Background] Smith-Bindman R, Chu PW, Ecker J, Feldstein VA, Filly RA, Bacchetti P. Adverse birth outcomes in relation to prenatal sonographic measurements of fetal size. J Ultrasound Med. 2003 Apr;22(4):347-56; quiz 357-8. doi: 10.7863/jum.2003.22.4.347. PMID 12693618
- [Background] Smith-Bindman R, Chu PW, Ecker JL, Feldstein VA, Filly RA, Bacchetti P. US evaluation of fetal growth: prediction of neonatal outcomes. Radiology. 2002 Apr;223(1):153-61. doi: 10.1148/radiol.2231010876. PMID 11930060
- [Background] Smith-Bindman R, Hosmer W, Feldstein VA, Deeks JJ, Goldberg JD. Second-trimester ultrasound to detect fetuses with Down syndrome: a meta-analysis. JAMA. 2001 Feb 28;285(8):1044-55. doi: 10.1001/jama.285.8.1044. PMID 11209176
- [Background] Smith-Bindman R, Hosmer WD, Caponigro M, Cunningham G. The variability in the interpretation of prenatal diagnostic ultrasound. Ultrasound Obstet Gynecol. 2001 Apr;17(4):326-32. doi: 10.1046/j.1469-0705.2001.00346.x. PMID 11339190
- [Background] Smith-Bindman R, Kerlikowske K, Feldstein VA, Subak L, Scheidler J, Segal M, Brand R, Grady D. Endovaginal ultrasound to exclude endometrial cancer and other endometrial abnormalities. JAMA. 1998 Nov 4;280(17):1510-7. doi: 10.1001/jama.280.17.1510. PMID 9809732
- [Background] Smith-Bindman R, Kerlikowske K, Gebretsadik T, Newman J. Is screening mammography effective in elderly women? Am J Med. 2000 Feb;108(2):112-9. doi: 10.1016/s0002-9343(99)00406-4. PMID 11126304
- [Background] Smith-Bindman R, McCulloch CE, Ding A, Quale C, Chu PW. Diagnostic imaging rates for head injury in the ED and states' medical malpractice tort reforms. Am J Emerg Med. 2011 Jul;29(6):656-64. doi: 10.1016/j.ajem.2010.01.038. Epub 2010 Jul 13. PMID 20630679
- [Background] Smith-Bindman R, Weiss E, Feldstein V. How thick is too thick? When endometrial thickness should prompt biopsy in postmenopausal women without vaginal bleeding. Ultrasound Obstet Gynecol. 2004 Oct;24(5):558-65. doi: 10.1002/uog.1704. PMID 15386607
- [Background] Stengel JW, Webb EM, Poder L, Yeh BM, Smith-Bindman R, Coakley FV. Acute appendicitis: clinical outcome in patients with an initial false-positive CT diagnosis. Radiology. 2010 Jul;256(1):119-26. doi: 10.1148/radiol.10091229. Epub 2010 May 26. PMID 20505066
- [Background] Venkatesan A, Chu P, Kerlikowske K, Sickles EA, Smith-Bindman R. Positive predictive value of specific mammographic findings according to reader and patient variables. Radiology. 2009 Mar;250(3):648-57. doi: 10.1148/radiol.2503080541. Epub 2009 Jan 21. PMID 19164116
- [Background] Goldstein RB, Bree RL, Benson CB, Benacerraf BR, Bloss JD, Carlos R, Fleischer AC, Goldstein SR, Hunt RB, Kurman RJ, Kurtz AB, Laing FC, Parsons AK, Smith-Bindman R, Walker J. Evaluation of the woman with postmenopausal bleeding: Society of Radiologists in Ultrasound-Sponsored Consensus Conference statement. J Ultrasound Med. 2001 Oct;20(10):1025-36. doi: 10.7863/jum.2001.20.10.1025. PMID 11587008
- [Background] Solberg LI, Vinz C, Trevis JE. A technology solution for the high-tech diagnostic imaging conundrum. Am J Manag Care. 2012 Aug;18(8):421-5. PMID 22928757
- [Background] Crain AL, Solberg LI, Unutzer J, Ohnsorg KA, Maciosek MV, Whitebird RR, Beck A, Molitor BA. Designing and implementing research on a statewide quality improvement initiative: the DIAMOND study and initiative. Med Care. 2013 Sep;51(9):e58-66. doi: 10.1097/MLR.0b013e318249d8a4. PMID 22322100
- [Background] Boyle R, Solberg L, Fiore M. Use of electronic health records to support smoking cessation. Cochrane Database Syst Rev. 2011 Dec 7;(12):CD008743. doi: 10.1002/14651858.CD008743.pub2. PMID 22161436
- [Background] Solberg LI. Care coordination: what is it, what are its effects and can it be sustained? Fam Pract. 2011 Oct;28(5):469-70. doi: 10.1093/fampra/cmr071. No abstract available. PMID 21926060
- [Background] Fontaine P, Flottemesch TJ, Solberg LI, Asche SE. Is consistent primary care within a patient-centered medical home related to utilization patterns and costs? J Ambul Care Manage. 2011 Jan-Mar;34(1):10-9. doi: 10.1097/JAC.0b013e3181ff7019. PMID 21160348
- [Background] Solberg LI, Glasgow RE, Unutzer J, Jaeckels N, Oftedahl G, Beck A, Maciosek MV, Crain AL. Partnership research: a practical trial design for evaluation of a natural experiment to improve depression care. Med Care. 2010 Jul;48(7):576-82. doi: 10.1097/MLR.0b013e3181dbea62. PMID 20508531
- [Background] Whitebird RR, Solberg LI, Margolis KL, Asche SE, Trangle MA, Wineman AP. Barriers to improving primary care of depression: perspectives of medical group leaders. Qual Health Res. 2013 Jun;23(6):805-14. doi: 10.1177/1049732313482399. Epub 2013 Mar 20. PMID 23515301
- [Background] Whitebird RR, Kreitzer M, Crain AL, Lewis BA, Hanson LR, Enstad CJ. Mindfulness-based stress reduction for family caregivers: a randomized controlled trial. Gerontologist. 2013 Aug;53(4):676-86. doi: 10.1093/geront/gns126. Epub 2012 Oct 15. PMID 23070934
- [Background] Jilcott S, Ammerman A, Sommers J, Glasgow RE. Applying the RE-AIM framework to assess the public health impact of policy change. Ann Behav Med. 2007 Oct;34(2):105-14. doi: 10.1007/BF02872666. PMID 17927550
- [Background] Whitebird RR, Kreitzer MJ, Lewis BA, Hanson LR, Crain AL, Enstad CJ, Mehta A. Recruiting and retaining family caregivers to a randomized controlled trial on mindfulness-based stress reduction. Contemp Clin Trials. 2011 Sep;32(5):654-61. doi: 10.1016/j.cct.2011.05.002. Epub 2011 May 12. PMID 21601010
- [Background] Whitebird RR, Kreitzer MJ, O'Connor PJ. Mindfulness-Based Stress Reduction and Diabetes. Diabetes Spectr. 2009 Sep 21;22(4):226-230. doi: 10.2337/diaspect.22.4.226. No abstract available. PMID 20657669
- [Background] Gaglio B, Shoup JA, Glasgow RE. The RE-AIM framework: a systematic review of use over time. Am J Public Health. 2013 Jun;103(6):e38-46. doi: 10.2105/AJPH.2013.301299. Epub 2013 Apr 18. PMID 23597377
- [Background] Boone JM, Hendee WR, McNitt-Gray MF, Seltzer SE. Radiation exposure from CT scans: how to close our knowledge gaps, monitor and safeguard exposure--proceedings and recommendations of the Radiation Dose Summit, sponsored by NIBIB, February 24-25, 2011. Radiology. 2012 Nov;265(2):544-54. doi: 10.1148/radiol.12112201. Epub 2012 Sep 10. PMID 22966066
- [Background] Boone JM. Method for evaluating bow tie filter angle-dependent attenuation in CT: theory and simulation results. Med Phys. 2010 Jan;37(1):40-8. doi: 10.1118/1.3264616. PMID 20175464
- [Background] Boone JM. Dose spread functions in computed tomography: a Monte Carlo study. Med Phys. 2009 Oct;36(10):4547-54. doi: 10.1118/1.3223634. PMID 19928086
- [Background] Huda W, Nickoloff EL, Boone JM. Overview of patient dosimetry in diagnostic radiology in the USA for the past 50 years. Med Phys. 2008 Dec;35(12):5713-28. doi: 10.1118/1.3013604. PMID 19175129
- [Background] Boone JM, Brunberg JA. Computed tomography use in a tertiary care university hospital. J Am Coll Radiol. 2008 Feb;5(2):132-8. doi: 10.1016/j.jacr.2007.07.008. PMID 18242530
- [Background] Boone JM. Multidetector CT: opportunities, challenges, and concerns associated with scanners with 64 or more detector rows. Radiology. 2006 Nov;241(2):334-7. doi: 10.1148/radiol.2412060169. No abstract available. PMID 17057062
- [Background] Boone JM, Kwan AL, Seibert JA, Shah N, Lindfors KK, Nelson TR. Technique factors and their relationship to radiation dose in pendant geometry breast CT. Med Phys. 2005 Dec;32(12):3767-76. doi: 10.1118/1.2128126. PMID 16475776
- [Background] Schindera ST, Nelson RC, Lee ER, Delong DM, Ngyen G, Toncheva G, Yoshizumi TT. Abdominal multislice CT for obese patients: effect on image quality and radiation dose in a phantom study. Acad Radiol. 2007 Apr;14(4):486-94. doi: 10.1016/j.acra.2007.01.030. PMID 17368219
- [Background] Schindera ST, Nelson RC, Toth TL, Nguyen GT, Toncheva GI, DeLong DM, Yoshizumi TT. Effect of patient size on radiation dose for abdominal MDCT with automatic tube current modulation: phantom study. AJR Am J Roentgenol. 2008 Feb;190(2):W100-5. doi: 10.2214/AJR.07.2891. PMID 18212190
- [Background] Szucs-Farkas Z, Kurmann L, Strautz T, Patak MA, Vock P, Schindera ST. Patient exposure and image quality of low-dose pulmonary computed tomography angiography: comparison of 100- and 80-kVp protocols. Invest Radiol. 2008 Dec;43(12):871-6. doi: 10.1097/RLI.0b013e3181875e86. PMID 19002059
- [Background] Schindera ST, Nelson RC, Yoshizumi T, Toncheva G, Nguyen G, DeLong DM, Szucs-Farkas Z. Effect of automatic tube current modulation on radiation dose and image quality for low tube voltage multidetector row CT angiography: phantom study. Acad Radiol. 2009 Aug;16(8):997-1002. doi: 10.1016/j.acra.2009.02.021. Epub 2009 May 5. PMID 19409820
- [Background] Szucs-Farkas Z, Schaller C, Bensler S, Patak MA, Vock P, Schindera ST. Detection of pulmonary emboli with CT angiography at reduced radiation exposure and contrast material volume: comparison of 80 kVp and 120 kVp protocols in a matched cohort. Invest Radiol. 2009 Dec;44(12):793-9. doi: 10.1097/RLI.0b013e3181bfe230. PMID 19884825
- [Background] Szucs-Farkas Z, Strautz T, Patak MA, Kurmann L, Vock P, Schindera ST. Is body weight the most appropriate criterion to select patients eligible for low-dose pulmonary CT angiography? Analysis of objective and subjective image quality at 80 kVp in 100 patients. Eur Radiol. 2009 Aug;19(8):1914-22. doi: 10.1007/s00330-009-1385-7. Epub 2009 Mar 31. PMID 19333605
- [Background] Marin D, Nelson RC, Schindera ST, Richard S, Youngblood RS, Yoshizumi TT, Samei E. Low-tube-voltage, high-tube-current multidetector abdominal CT: improved image quality and decreased radiation dose with adaptive statistical iterative reconstruction algorithm--initial clinical experience. Radiology. 2010 Jan;254(1):145-53. doi: 10.1148/radiol.09090094. PMID 20032149
- [Background] Schindera ST, Nauer C, Treier R, Trueb P, von Allmen G, Vock P, Szucs-Farkas Z. [Strategies for reducing the CT radiation dose]. Radiologe. 2010 Dec;50(12):1120, 1122-7. doi: 10.1007/s00117-010-2053-2. German. PMID 20844858
- [Background] Marin D, Nelson RC, Guerrisi A, Barnhart H, Schindera ST, Passariello R, Catalano C. 64-section multidetector CT of the upper abdomen: optimization of a saline chaser injection protocol for improved vascular and parenchymal contrast enhancement. Eur Radiol. 2011 Sep;21(9):1938-47. doi: 10.1007/s00330-011-2139-x. Epub 2011 May 11. PMID 21556911
- [Background] Marin D, Nelson RC, Rubin GD, Schindera ST. Body CT: technical advances for improving safety. AJR Am J Roentgenol. 2011 Jul;197(1):33-41. doi: 10.2214/AJR.11.6755. PMID 21701008
- [Background] Schindera ST, Diedrichsen L, Muller HC, Rusch O, Marin D, Schmidt B, Raupach R, Vock P, Szucs-Farkas Z. Iterative reconstruction algorithm for abdominal multidetector CT at different tube voltages: assessment of diagnostic accuracy, image quality, and radiation dose in a phantom study. Radiology. 2011 Aug;260(2):454-62. doi: 10.1148/radiol.11102217. Epub 2011 Apr 14. PMID 21493795
- [Background] Szucs-Farkas Z, Schibler F, Cullmann J, Torrente JC, Patak MA, Raible S, Hoppe H, Wyttenbach R, Vock P, Schindera ST. Diagnostic accuracy of pulmonary CT angiography at low tube voltage: intraindividual comparison of a normal-dose protocol at 120 kVp and a low-dose protocol at 80 kVp using reduced amount of contrast medium in a simulation study. AJR Am J Roentgenol. 2011 Nov;197(5):W852-9. doi: 10.2214/AJR.11.6750. PMID 22021532
- [Background] Schindera ST, Odedra D, Raza SA, Kim TK, Jang HJ, Szucs-Farkas Z, Rogalla P. Iterative reconstruction algorithm for CT: can radiation dose be decreased while low-contrast detectability is preserved? Radiology. 2013 Nov;269(2):511-8. doi: 10.1148/radiol.13122349. Epub 2013 Jun 20. PMID 23788715
- [Background] Loupatatzis C, Schindera S, Gralla J, Hoppe H, Bittner J, Schroder R, Srivastav S, Bonel HM. Whole-body computed tomography for multiple traumas using a triphasic injection protocol. Eur Radiol. 2008 Jun;18(6):1206-14. doi: 10.1007/s00330-008-0875-3. Epub 2008 Feb 13. PMID 18270712
- [Background] Solberg L. Quality improvement in primary care: The role of organization, systems, and collaboratives. In: Sollecito WA, Johnson JK, eds. McLaughlin and Kaluzny's continuous quality improvement in health care. Fourth ed. Burlington, MA: Jones & Bartlett Learning; 399-419. 2011
- [Background] Solberg LI, Brekke ML, Fazio CJ, Fowles J, Jacobsen DN, Kottke TE, Mosser G, O'Connor PJ, Ohnsorg KA, Rolnick SJ. Lessons from experienced guideline implementers: attend to many factors and use multiple strategies. Jt Comm J Qual Improv. 2000 Apr;26(4):171-88. doi: 10.1016/s1070-3241(00)26013-6. PMID 10749003
- [Background] Solberg LI, Kottke TE, Brekke ML, Magnan S. Improving prevention is difficult. Eff Clin Pract. 2000 May-Jun;3(3):153-5. No abstract available. PMID 11182966
- [Background] Solberg LI, Hroscikoski MC, Sperl-Hillen JM, O'Connor PJ, Crabtree BF. Key issues in transforming health care organizations for quality: the case of advanced access. Jt Comm J Qual Saf. 2004 Jan;30(1):15-24. doi: 10.1016/s1549-3741(04)30002-x. PMID 14738032
- [Background] Hroscikoski MC, Solberg LI, Sperl-Hillen JM, Harper PG, McGrail MP, Crabtree BF. Challenges of change: a qualitative study of chronic care model implementation. Ann Fam Med. 2006 Jul-Aug;4(4):317-26. doi: 10.1370/afm.570. PMID 16868235
- [Background] Solberg LI, Crain AL, Sperl-Hillen JM, Hroscikoski MC, Engebretson KI, O'Connor PJ. Care quality and implementation of the chronic care model: a quantitative study. Ann Fam Med. 2006 Jul-Aug;4(4):310-6. doi: 10.1370/afm.571. PMID 16868234
- [Background] Solberg LI, Engebretson KI, Sperl-Hillen JM, O'Connor PJ, Hroscikoski MC, Crain AL. Ambulatory care quality measures for the 6 aims from administrative data. Am J Med Qual. 2006 Sep-Oct;21(5):310-6. doi: 10.1177/1062860606289071. PMID 16973947
- [Background] Solberg LI, Taylor N, Conway WA, Hiatt RA. Large multispecialty group practices and quality improvement: what is needed to transform care? J Ambul Care Manage. 2007 Jan-Mar;30(1):9-17; discussion 18-20. doi: 10.1097/00004479-200701000-00003. PMID 17170633
- [Background] American Association of Physicists in Medicine Position Statement on Radiation Risks from Medical Imaging Procedures. 2011
- [Background] Huda W, Magill D, He W. CT effective dose per dose length product using ICRP 103 weighting factors. Med Phys. 2011 Mar;38(3):1261-5. doi: 10.1118/1.3544350. PMID 21520838
- [Background] The 2007 Recommendations of the International Commission on Radiological Protection. ICRP publication 103. Ann ICRP. 2007;37(2-4):1-332. doi: 10.1016/j.icrp.2007.10.003. PMID 18082557
- [Background] Land CE. Studies of cancer and radiation dose among atomic bomb survivors. The example of breast cancer. JAMA. 1995 Aug 2;274(5):402-7. PMID 7616636
- [Background] Linet MS, Kim KP, Rajaraman P. Children's exposure to diagnostic medical radiation and cancer risk: epidemiologic and dosimetric considerations. Pediatr Radiol. 2009 Feb;39 Suppl 1(Suppl 1):S4-26. doi: 10.1007/s00247-008-1026-3. Epub 2008 Dec 16. PMID 19083224
- [Background] Brenner D, Elliston C, Hall E, Berdon W. Estimated risks of radiation-induced fatal cancer from pediatric CT. AJR Am J Roentgenol. 2001 Feb;176(2):289-96. doi: 10.2214/ajr.176.2.1760289. PMID 11159059
- [Background] Feigal DW Jr. FDA public health notification: reducing radiation risk from computed tomography for pediatric and small adult patients. Int J Trauma Nurs. 2002 Jan-Mar;8(1):1-2. doi: 10.1067/mtn.2002.121511. No abstract available. PMID 11793002
- [Background] Brenner DJ, Hall EJ. Computed tomography--an increasing source of radiation exposure. N Engl J Med. 2007 Nov 29;357(22):2277-84. doi: 10.1056/NEJMra072149. No abstract available. PMID 18046031
- [Background] National Research Council (US) Committee on the Biological Effects of Ionizing Radiation (BEIR V). Health Effects of Exposure to Low Levels of Ionizing Radiation: Beir V. Washington (DC): National Academies Press (US); 1990. Available from http://www.ncbi.nlm.nih.gov/books/NBK218704/ PMID 25032334
- [Background] Paterson A, Frush DP, Donnelly LF. Helical CT of the body: are settings adjusted for pediatric patients? AJR Am J Roentgenol. 2001 Feb;176(2):297-301. doi: 10.2214/ajr.176.2.1760297. PMID 11159060
- [Background] American Association of Physicists in Medicine. AAPM Report No 96. The Measurement, reporting and management of radiation dose in CT, Report of AAPM Task group 23 of the Diagnostic Imaging Council CT Committee. College Park, MD: American Association of Physicists in Medicine; 2008
- [Background] NQF. National Quality Forum Measure 0739, Radiation Dose of Computed Tomography (CT) Steward: University of California San Francisco. 2011; http://www.qualityforum.org/QPS/0739
- [Background] Mittman B. Implementation Science in Health Care. In: Brownson RC, Colditz GA, Proctor EK, eds. Dissemination and Implementation Research in Health. New York: Oxford University Press; 2012:400-418
- [Background] Solberg LI. Guideline implementation: what the literature doesn't tell us. Jt Comm J Qual Improv. 2000 Sep;26(9):525-37. doi: 10.1016/s1070-3241(00)26044-6. PMID 10983293
- [Background] Chaillet N, Dube E, Dugas M, Audibert F, Tourigny C, Fraser WD, Dumont A. Evidence-based strategies for implementing guidelines in obstetrics: a systematic review. Obstet Gynecol. 2006 Nov;108(5):1234-45. doi: 10.1097/01.AOG.0000236434.74160.8b. PMID 17077251
- [Background] Jamtvedt G, Young JM, Kristoffersen DT, O'Brien MA, Oxman AD. Does telling people what they have been doing change what they do? A systematic review of the effects of audit and feedback. Qual Saf Health Care. 2006 Dec;15(6):433-6. doi: 10.1136/qshc.2006.018549. PMID 17142594
- [Background] Shojania KG, Ranji SR, McDonald KM, Grimshaw JM, Sundaram V, Rushakoff RJ, Owens DK. Effects of quality improvement strategies for type 2 diabetes on glycemic control: a meta-regression analysis. JAMA. 2006 Jul 26;296(4):427-40. doi: 10.1001/jama.296.4.427. PMID 16868301
- [Background] Prior M, Guerin M, Grimmer-Somers K. The effectiveness of clinical guideline implementation strategies--a synthesis of systematic review findings. J Eval Clin Pract. 2008 Oct;14(5):888-97. doi: 10.1111/j.1365-2753.2008.01014.x. PMID 19018923
- [Background] Hysong SJ. Meta-analysis: audit and feedback features impact effectiveness on care quality. Med Care. 2009 Mar;47(3):356-63. doi: 10.1097/MLR.0b013e3181893f6b. PMID 19194332
- [Background] Grimshaw J, Eccles M, Thomas R, MacLennan G, Ramsay C, Fraser C, Vale L. Toward evidence-based quality improvement. Evidence (and its limitations) of the effectiveness of guideline dissemination and implementation strategies 1966-1998. J Gen Intern Med. 2006 Feb;21 Suppl 2(Suppl 2):S14-20. doi: 10.1111/j.1525-1497.2006.00357.x. PMID 16637955
- [Background] Brown CA, Lilford RJ. The stepped wedge trial design: a systematic review. BMC Med Res Methodol. 2006 Nov 8;6:54. doi: 10.1186/1471-2288-6-54. PMID 17092344
- [Background] Stone EG, Morton SC, Hulscher ME, Maglione MA, Roth EA, Grimshaw JM, Mittman BS, Rubenstein LV, Rubenstein LZ, Shekelle PG. Interventions that increase use of adult immunization and cancer screening services: a meta-analysis. Ann Intern Med. 2002 May 7;136(9):641-51. doi: 10.7326/0003-4819-136-9-200205070-00006. PMID 11992299
- [Background] Leconte I, Feger C, Galant C, Berliere M, Berg BV, D'Hoore W, Maldague B. Mammography and subsequent whole-breast sonography of nonpalpable breast cancers: the importance of radiologic breast density. AJR Am J Roentgenol. 2003 Jun;180(6):1675-9. doi: 10.2214/ajr.180.6.1801675. PMID 12760942
- [Background] Marshall C, & Rossman, G.B. Designing Qualitative Research. 4th ed. Newbury Park: Sage Publications; 2006.
- [Background] Huberman MM. Qualitative Data Analysis: An Expanded Sourcebook. Thousand Oaks, CA: Sage Publications; 1994.
- [Background] Patton MQ. Qualitative Research and Evaluation Methods. 3rd ed. Newbury Park: Sage Publications; 2002.
- [Background] Padgett D. Qualitative Methods in Social Work Research: Challenges and Rewards. Thousand Oaks, CA: Sage; 1998
- [Background] Seale C. The Quality of Qualitative Research. Thousand Oaks: Sage Publications; 1999
- [Background] Greevy R, Lu B, Silber JH, Rosenbaum P. Optimal multivariate matching before randomization. Biostatistics. 2004 Apr;5(2):263-75. doi: 10.1093/biostatistics/5.2.263. PMID 15054030
- [Background] Greevy RA Jr, Grijalva CG, Roumie CL, Beck C, Hung AM, Murff HJ, Liu X, Griffin MR. Reweighted Mahalanobis distance matching for cluster-randomized trials with missing data. Pharmacoepidemiol Drug Saf. 2012 May;21 Suppl 2(0 2):148-54. doi: 10.1002/pds.3260. PMID 22552990
- [Background] 171. Morgan KL, Rubin, D.L. Rerandomization to improve covariate balance in experiments. The Annals of Statistics 2012;40:1263-82.
- [Result] Smith-Bindman R, Chu P, Wang Y, Chung R, Lopez-Solano N, Einstein AJ, Solberg L, Cervantes LF, Yellen-Nelson T, Boswell W, Delman BN, Duong PA, Goode AR, Kasraie N, Lee RK, Neill R, Pahwa A, Pike P, Roehm J, Schindera S, Starkey J, Suntharalingam S, Jeukens CRLPN, Miglioretti DL. Comparison of the Effectiveness of Single-Component and Multicomponent Interventions for Reducing Radiation Doses in Patients Undergoing Computed Tomography: A Randomized Clinical Trial. JAMA Intern Med. 2020 May 1;180(5):666-675. doi: 10.1001/jamainternmed.2020.0064. PMID 32227142
- [Derived] Smith-Bindman R, Wang Y, Chu P, Chung R, Einstein AJ, Balcombe J, Cocker M, Das M, Delman BN, Flynn M, Gould R, Lee RK, Nelson TR, Schindera S, Seibert A, Starkey J, Suntharalingam S, Wetter A, Wildberger JE, Miglioretti DL. International variation in radiation dose for computed tomography examinations: prospective cohort study. BMJ. 2019 Jan 2;364:k4931. doi: 10.1136/bmj.k4931. PMID 30602590
- See also: The website explores and focuses on studying the impact of medical imaging on health, minimizing the harms of medical imaging and and providing rigorous evidence to aid policymakers regarding use of medical imaging. — http://ctdose.ucsf.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study subjects were passively enrolled in this study; we had a waiver of informed consent and there was no direct contact with subjects. We have listed the number of unique subjects enrolled into each track; however, ALL ANALYSES WERE PERFORMED AT THE LEVEL OF THE CT SCAN, not at the individual subject level.
Units Other Than Participants: CT scans
Groups:
- Track A: Track A received the simple audit intervention at week 40 and the multi-component intervention at week 68.
  The simple audit provided feedback on radiation doses including comparison with other participating sites. The multi-component intervention gave tailored, actionable feedback on needed changes in addition to a 7-week quality improvement collaborative that included guidance on quality improvement methods, webinars, interactive lectures by experts, case reviews, and best practices sharing.
- Track B: Track B received the simple audit intervention at week 44 and the multi-component intervention at week 74.
  The simple audit provided feedback on radiation doses including comparison with other participating sites. The multi-component intervention gave tailored, actionable feedback on needed changes in addition to a 7-week quality improvement collaborative that included guidance on quality improvement methods, webinars, interactive lectures by experts, case reviews, and best practices sharing.
- Track C: Track C received the simple audit intervention at week 53 and the multi-component intervention at week 81.
  The simple audit provided feedback on radiation doses including comparison with other participating sites. The multi-component intervention gave tailored, actionable feedback on needed changes in addition to a 7-week quality improvement collaborative that included guidance on quality improvement methods, webinars, interactive lectures by experts, case reviews, and best practices sharing.
Period: Overall Study
Arm/Group | Track A | Track B | Track C
Started | 251607; 327,462 CT scans (Track A Imaging facilities: 32) | 229022; 306,825 CT scans (Track B Imaging facilities: 29) | 383451; 522,370 CT scans (Track C Imaging facilities: 39)
Completed (All subjects started and completed each track. Note, however, that patients were enrolled passively. The unit of analysis was CT scans (not individual subjects), and all eligible CT scans performed during each study period were included.) | 251607; 327,462 CT scans | 229022; 306,825 CT scans | 383451; 522,370 CT scans
Not Completed | 0; NA CT scans | 0; NA CT scans | 0; NA CT scans

BASELINE CHARACTERISTICS:
Population: THE UNIT OF ANALYSIS IS CT SCANS, NOT PATIENTS. The arms in this section do not reflect the randomization tracks (A,B,C) but rather study periods: before intervention; after simple audit; after multi-component intervention. We excluded scans obtained during transition ("washout") periods immediately following each intervention. The numbers here reflect unique CT scans, not unique patients. Units are not counted more than once.
Units Other Than Participants: CT scans
Groups:
- Baseline Period: Reflects CT scans analyzed during a baseline period of usual care (before intervention). The duration of this period differed by randomization Track (A, B, or C).
- Simple Audit Intervention Period: Reflects CT scans analyzed after receiving the simple audit report intervention. The duration of this period differed by randomization Track (A, B, or C).
- Multi-component Intervention Period: Reflects CT scans analyzed after receiving the multi-component intervention. The duration of this period differed by randomization Track (A, B, or C).
- Total: Total of all reporting groups
Arm/Group | Baseline Period | Simple Audit Intervention Period | Multi-component Intervention Period | Total
Number analyzed (Participants) | NA | NA | NA | NA
Number analyzed (CT scans) | 526439 | 251409 | 207576 | 985424
Age, Customized [Count of Units; unit: CT scans] — Patient age distribution by decade.
  CT scans
    18-29 years | 40022 | 18468 | 15391 | 73881
    30-39 years | 45880 | 21198 | 17615 | 84693
    40-49 years | 64299 | 29492 | 24351 | 118142
    50-59 years | 98457 | 46589 | 37951 | 182997
    60-69 years | 114161 | 54155 | 44102 | 212418
    70-79 years | 92374 | 45969 | 39073 | 177416
    80 years and older | 71246 | 35538 | 29093 | 135877
Sex: Female, Male [Count of Units; unit: CT scans]
  Female | 278841 | 132772 | 110088 | 521701
  Male | 247598 | 118637 | 97488 | 463723
Ethnicity (NIH/OMB) [Count of Units; unit: CT scans] — Race and Ethnicity data not collected
  CT scans
    Hispanic or Latino | NA — Race and Ethnicity data not collected | NA — Race and Ethnicity data not collected | NA — Race and Ethnicity data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
    Not Hispanic or Latino | NA — Race and Ethnicity data not collected | NA — Race and Ethnicity data not collected | NA — Race and Ethnicity data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
    Unknown or Not Reported | NA — Race and Ethnicity data not collected | NA — Race and Ethnicity data not collected | NA — Race and Ethnicity data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
Race (NIH/OMB) [Count of Units; unit: CT scans] — Race and Ethnicity data not collected
  CT scans
    American Indian or Alaska Native | NA — Race and Ethnicity data not collected | NA — Race and Ethnicity data not collected | NA — Race and Ethnicity data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
    Asian | NA — Race and Ethnicity data not collected | NA — Race and Ethnicity data not collected | NA — Race and Ethnicity data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
    Native Hawaiian or Other Pacific Islander | NA — Race and Ethnicity data not collected | NA — Race and Ethnicity data not collected | NA — Race and Ethnicity data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
    Black or African American | NA — Race and Ethnicity data not collected | NA — Race and Ethnicity data not collected | NA — Race and Ethnicity data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
    White | NA — Race and Ethnicity data not collected | NA — Race and Ethnicity data not collected | NA — Race and Ethnicity data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
    More than one race | NA — Race and Ethnicity data not collected | NA — Race and Ethnicity data not collected | NA — Race and Ethnicity data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
    Unknown or Not Reported | NA — Race and Ethnicity data not collected | NA — Race and Ethnicity data not collected | NA — Race and Ethnicity data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
Type of scan [Count of Units; unit: CT scans] — Anatomical region imaged.
  CT scans
    Abdomen | 185671 | 87518 | 72084 | 345273
    Chest | 143120 | 69678 | 56410 | 269208
    Combined abdomen and chest | 30689 | 14784 | 14416 | 59889
    Head | 166959 | 79429 | 64666 | 311054
Age, by type of scan [Mean (Standard Deviation); unit: Years]
  Abdomen | 56.0 (18.2) | 56.3 (18.3) | 56.4 (18.3) | 56.2 (18.3)
  Chest | 61.6 (15.3) | 62.1 (15.2) | 62.0 (15.2) | 61.8 (15.2)
  Combined abdomen and chest | 62.5 (15.3) | 62.8 (15.5) | 63.4 (15.4) | 62.8 (15.4)
  Head | 60.1 (19.9) | 60.7 (19.9) | 60.6 (19.9) | 60.4 (19.9)
Patient diameter [Mean (Standard Deviation); unit: Centimeters (cm)] — Patient diameter, as measured in cm on mid-scan images, is an indicator of patient size.
  Centimeters (cm)
    Abdomen | 30.7 (4.6) | 30.8 (4.7) | 30.9 (4.7) | 30.8 (4.7)
    Chest | 28.9 (4.9) | 29.0 (4.9) | 28.9 (5.1) | 28.9 (5.0)
    Combined abdomen and chest | 29.7 (4.1) | 29.5 (4.2) | 29.7 (4.2) | 29.7 (4.2)
    Head | 17.1 (1.5) | 17.1 (1.5) | 17.2 (1.5) | 17.1 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Effective Dose (ED)
Description: We will assess the change in the mean effective dose after the simple audit and multi-component interventions (MCI) in comparison to before the audit and multi-component interventions. The numbers given below reflect absolute change in mean dose (in millisieverts) relative to the baseline period.
Time Frame: Sites were randomized to 1 of 3 tracks, which determined the timing of intervention: Track A: audit at week 40, MCI at week 68 Track B: audit at week 44, MCI at week 74 Track C: audit at week 53, MCI at week 81
Population: The unit of analysis is CT scans; there were no data collected at the participant level. We excluded scans obtained during transition ("washout") periods immediately following each intervention. The numbers given below reflect absolute change in mean dose (in millisieverts) relative to the baseline period.
Measure: Mean (95% Confidence Interval); unit: Millisieverts (mSv)
Units Other Than Participants: CT scans
Groups:
- Simple Audit Intervention Period: Reflects CT scans analyzed after receiving the simple audit report intervention.
- Multi-component Intervention Period: Reflects CT scans analyzed after receiving the multi-component intervention.
Arm/Group | Simple Audit Intervention Period | Multi-component Intervention Period
Number analyzed (Participants) | NA | NA
Number analyzed (CT scans) | 251409 | 207576
Millisieverts (mSv)
  Abdomen | -0.13 [-0.24 to -0.02] | -0.81 [-0.99 to -0.64]
  Chest | -0.14 [-0.23 to -0.05] | -0.26 [-0.40 to -0.11]
  Combined abdomen and chest | -0.88 [-1.18 to -0.57] | -2.04 [-2.55 to -1.53]
  Head | -0.01 [-0.06 to 0.04] | -0.05 [-0.13 to 0.02]

2. Primary Outcome: Percentage of CT Scans With an Effective Dose Above Benchmark
Description: We will assess the change in the percentage of examinations with an effective dose above the benchmark after the simple audit and after multi-component intervention (MCI) in comparison to doses before the audit and MCI. The benchmark for each anatomic area is defined as the 75th percentile of the dose distribution during the pre-intervention (baseline) period.
Time Frame: as for outcome 1
Population: The unit of analysis is CT scans; there were no data collected at the participant level. We excluded scans obtained during transition ("washout") periods immediately following each intervention.
Measure: Number; unit: Percent of CT scans over benchmark
Units Other Than Participants: CT scans
Groups:
- Baseline Period: Reflects CT scans analyzed during a baseline period of usual care (before intervention).
Arm/Group | Baseline Period | Simple Audit Intervention Period | Multi-component Intervention Period
Number analyzed (Participants) | NA | NA | NA
Number analyzed (CT scans) | 526439 | 251409 | 207576
Percent of CT scans over benchmark
  Abdomen | 24.7 | 24.7 | 22.2
  Chest | 26 | 25.5 | 24.9
  Combined chest and abdomen | 26.7 | 23 | 18.8
  Head | 26.2 | 26 | 21.8

3. Secondary Outcome: Mean Dose Length Product
Description: We will assess the change in the dose length product after the audit and MCI in comparison to before the audit and MCI.
Time Frame: as for outcome 1
Population: Data were not collected.
Arm/Group | Baseline Period | Simple Audit Intervention Period | Multi-component Intervention Period
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Proportion of CT Scans With a Dose Length Product Above Benchmark
Description: We will assess the change in the proportion of examinations with a dose length product above the benchmark after the audit and after the MCI in comparison to doses before the audit and MCI. The benchmark for each anatomic area is defined as the 75th percentile of the dose distribution during the pre intervention period.
Time Frame: as for outcome 1
Population: Data were not collected.
Arm/Group | Baseline Period | Simple Audit Intervention Period | Multi-component Intervention Period
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Change in Mean Volume Computed Tomography Dose Index (CTDIvol)
Description: We will assess the change in the mean volume CT dose index (CTDIvol) from before versus after the audit and MCI intervention. CTDIvol (in units of milligray, mGy) is a measure of radiation dose, reflecting the amount of radiation imparted per CT slice by the scanner. Higher CTDIvol signifies more radiation dose. In general, a reduction in CTDIvol would be a sign of quality improvement, minimizing excess radiation exposure to the patient.
Time Frame: as for outcome 1
Population: The unit of analysis is CT scans; there were no data collected at the participant level. We excluded scans obtained during transition ("washout") periods immediately following each intervention. The numbers given below reflect absolute change in mean dose (in milligray, mGy) relative to the baseline period.
Measure: Mean (95% Confidence Interval); unit: Milligrays (mGy)
Units Other Than Participants: CT scans
Arm/Group | Simple Audit Intervention Period | Multi-component Intervention Period
Number analyzed (Participants) | NA | NA
Number analyzed (CT scans) | 251409 | 207576
Milligrays (mGy)
  Abdomen | 0.09 [0.01 to 0.16] | 0.03 [-0.10 to 0.15]
  Chest | 0.04 [-0.07 to 0.14] | -0.11 [-0.29 to 0.06]
  Combined abdomen and chest | -0.05 [-0.18 to 0.08] | -0.42 [-0.64 to -0.20]
  Head | 0.44 [0.27 to 0.62] | -0.56 [-0.85 to -0.27]

6. Secondary Outcome: Percentage of CT Scans With a CTDIvol Above Benchmark
Description: We will assess the change in the percentage of examinations with a CTDIvol above the benchmark after the audit and after multicomponent intervention in comparison to doses before the audit and multicomponent intervention. The benchmark for each anatomic area is defined as the 75th percentile of the dose distribution during the pre intervention period.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: Percentage of CT scans
Units Other Than Participants: CT scans
Arm/Group | Baseline Period | Simple Audit Intervention Period | Multi-component Intervention Period
Number analyzed (Participants) | NA | NA | NA
Number analyzed (CT scans) | 526439 | 251409 | 207576
Percentage of CT scans
  Abdomen | 24.5 | 24.9 | 24.1
  Chest | 26 | 25.8 | 24.1
  Combined chest and abdomen | 23.6 | 22.7 | 19.9
  Head | 24.4 | 25.0 | 17.9

7. Secondary Outcome: Change in Mean Organ Doses: Brain Dose for Head CT; Lung Dose For Chest CT; Colon and Liver Dose for Abdomen CT
Description: We will assess the change in organ doses after the simple audit and multi-component interventions (MCI) in comparison to before the audit and multi-component interventions. The numbers given below reflect absolute change in mean dose (in millisieverts) relative to the baseline period.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Milligrays (mGy)
Units Other Than Participants: CT scans
Arm/Group | Simple Audit Intervention Period | Multi-component Intervention Period
Number analyzed (Participants) | NA | NA
Number analyzed (CT scans) | 251409 | 207576
Milligrays (mGy)
  Abdomen (colon organ dose) | -6.0 [-6.9 to -5.0] | -12.2 [-13.8 to -10.6]
  Chest (lung organ dose) | -2.1 [-2.8 to -1.5] | -3.7 [-4.7 to -2.7]
  Combined chest and abdomen (lung organ dose) | -16.0 [-18.2 to -13.8] | -30.1 [-33.8 to -26.4]
  Combined chest and abdomen (colon organ dose) | -13.0 [-14.5 to -11.6] | -17.6 [-20.0 to -15.1]
  Head (brain organ dose) | -2.9 [-6.4 to 0.70] | -7.5 [-13.3 to -1.7]

ADVERSE EVENTS:
Time Frame: Adverse events were not collected.
Description: Adverse event data were not reported in this study. Study data were collected from consecutive patients who underwent a standard of care procedure (CT imaging). No tests, treatments, or interactions with any patients were performed as part of this study. There was no way to capture, nor any need to capture for the purpose of our research, adverse events related to their imaging procedures.
Groups:
- Track A; Track B: Simple Audit Report In-Person Meeting Multi-Component Intervention
  Simple Audit Report: The simple audit provides comparison and feedback on radiation doses.
  Multi-Component Intervention: The multi-component intervention gives tailored feedback on needed changes plus guidance using quality improvement methods that facilitate organizational change. Provides access to experts, detailed audit, collaborative calls, and site visits (as needed).
  In-Person Meeting: Collaborator meeting with an emphasis on quality improvement.
- Track C: Simple Audit Report Multi-Component Intervention
  Simple Audit Report: The simple audit provides comparison and feedback on radiation doses.
  Multi-Component Intervention: The multi-component intervention gives tailored feedback on needed changes plus guidance using quality improvement methods that facilitate organizational change. Provides access to experts, detailed audit, collaborative calls, and site visits (as needed).
Arm/Group | Track A | Track B | Track C
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT03000751/Prot_SAP_002.pdf